CLINICAL TRIAL: NCT06156644
Title: Pulsed-Field-Ablation to Treat Atrial fiBRillation With a novEl multimodalIty Generator
Acronym: PFA-Breisgau
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, PD Dr. Dirk Westermann, Prof, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PFA-Breisgau
Record Dates: First submitted 2023-11-13; First posted 2023-12-05 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Single Arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PFA strategy (Other): PFA will be performed based on a specific protocol
  Interventions: Device: PFA

INTERVENTIONS:
Device: PFA — Ablation to treat trail fibrillation

SUMMARY:
In this first-in-human clinical trial a novel generator (INTELLAPULSE), designed and built by Stockert, which supports highly flexible PFA protocols as well as RF interventions will be used. For 12 months and follow-up for 12 months, after a 3-months blanking period 50 consecutive paroxysmal AF patients, eligible for catheter ablation, will be enrolled.

DETAILED DESCRIPTION:
The principal safety and efficacy of PFA have been established in previous studies, showing low compli¬cation rates, short procedure times, and non-inferior/ superior efficiency compared to thermal abla¬tion.18, 19 However, current generators available for clinical practice are not generally designed to allow both non-thermal and thermal ablation in single shot settings. Moreover, modification of PFA sequences is not supported in commercially available systems. Flexible, multi-modal generators that allow one to conduct PFA or RF ablation using one and the same catheter would be highly desirable, from a clinical point of view, to allow for on-the-fly decision-making in view of individual patient requirements.

In this first-in-human clinical trial a novel generator (INTELLAPULSE), designed and built by Stockert, which supports highly flexible PFA protocols as well as RF interventions will be used. This generator will be CE marked in Q3/24. Upon completion of the ethical approval process in Q2/25, the 'first in human' study, exploring safety of the Stockert PFA generator will be started.

The trial will be a prospective single arm study at the UHZ Freiburg · Bad Krozingen and will recruit for 12 months and follow-up for 12 months, after a 3-months blanking period. 50 consecutive paroxysmal AF patients, eligible for catheter ablation, will be enrolled. Exclusion criteria will be age <18 years, previous left atrial ablation, and lack or withdrawal of written informed consent. Data acquisition will use an electronic case report form (RedCap Database). Procedures will be performed using standard operating procedures (SOP).

In short: ablations will be performed under deep analgo-sedation and/or general anaesthesia. Trans¬oesophageal echocardiography will be performed if patients present with either AF or atrial tachycardia (to exclude intracardiac thrombi) or in sinus rhythm (in patients with interrupted oral anticoagulation and CHA2DS2-VASc-Score ≥2). Atrial transseptal puncture will be performed for access to pulmonary veins (PV), using a fixed curve transseptal sheath and transseptal needle according to standard SOP. PFA catheters (FARAWAVE™, Boston Scientific) will be utilized, as in prior work with a commercial PFA system (FARAPULSE™, Boston Scientific) at the UHZ. At every PV antrum, 8 PFA-pulses will be delivered in 'flower' and 'basket' configurations (delivery of additional PFA-pulses will be at operator's discretion).

ELIGIBILITY:
Inclusion Criteria:

* new onset atrial fibrillation

Exclusion Criteria:

* age <18 years
* previous left atrial ablation
* lack or withdrawal of written informed consent
* unable to receive ablation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
number of death | 12 month
  Primary endpoints focusing of the safety of the strategy

IPD SHARING:
Plan to Share IPD: No